CLINICAL TRIAL: NCT02498080
Title: Drug Eluting Balloons Versus Standard Percutaneous Transluminal Angioplasty in Infra-popliteal Arteries in Patients With Critical Limb Ischemia: a Randomized Clinical Trial
Brief Title: Drug Eluting Balloons PTA in Infra-popliteal Arteries in Patients With Critical Limb Ischemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Francesco Pompeo, Head of vascular surgery division, Neuromed IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pmp01
Record Dates: First submitted 2015-07-06; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Critical Limb Ischemia
Keywords: Drug eluting balloons; Critical limb ischemia; Infra-popliteal arteries; Percutaneous transluminal angioplasty
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DEB PTA (Experimental): Devices: paclitaxel drug eluting balloon PTA
  Interventions: Procedure: DEB PTA
- standard PTA (Active Comparator): devices: standard balloon PTA
  Interventions: Procedure: Standard PTA

INTERVENTIONS:
Procedure: DEB PTA — paclitaxel drug eluting balloon PTA
  Arms: DEB PTA
Procedure: Standard PTA — Standard PTA
  Arms: standard PTA

SUMMARY:
Percutaneous transluminal angioplasty (PTA) of infra-popliteal arteries in patients suffering peripheral arterial occlusive disease (PAOD) provides good results in terms of limb salvage. During the last decade, drug eluting balloons (DEB) were found to be an effective tool for the treatment of atherosclerotic disease in several arterial districts. Aim of this study is to compare results of DEB PTA versus standard PTA of infra-popliteal district in patients with CLI, from a single-centre prospective randomized trial.

DETAILED DESCRIPTION:
Percutaneous transluminal angioplasty (PTA) of infra-popliteal arteries in patients suffering peripheral arterial occlusive disease (PAOD) provides good results in terms of limb salvage. Nevertheless, this treatment is still burdened by consistent restenosis and reintervention rates up to 68% and 50%, respectively.

During the last decade, drug eluting balloons (DEB) were found to be an effective tool for the treatment of atherosclerotic disease in several arterial districts. DEBs are coated by antimitotic drug (usually paclitaxel) in order to inhibit endothelial cells proliferation. Paclitaxel effectiveness is due to the drug lipophilicity.

A short (1 to 3 minutes) balloon inflation at the target vessel level is sufficient to deliver a therapeutic dose of paclitaxel, lasting in situ thereafter for months.

The effectiveness of DEBs has been already proven in coronary as well as in femoro-popliteal district: DEBs have improved primary patency rates both in de novo lesions and in femoro-popliteal intrastent restenosis.

A role for DEBs in the treatment of infra-popliteal lesions district in patients with critical limb ischemia (CLI) has been also described, however results in that specific anatomical site are still controversial.

The DEBATE-BTK Trial showed that DEBs reduce 1-year restenosis, target lesions revascularization (TLR) and target vessel occlusions rates in the treatment of infra-popliteal lesions in diabetic patients with CLI, compared with standard PTA. On the other hand, the IN.PACT DEEP Trial showed a higher major amputation rate and lower amputation-free survival for DEB compared to standard PTA.

It has been hypothesized that DEBs failure could be related to different materials and drug coating process for older DEBs, resulting in an insufficient dose delivered to the target vessel wall.

Aim of this study is to compare results of DEB PTA versus standard PTA of infra-popliteal district in patients with CLI, from a single-centre prospective randomized trial.

Patients and Methods

Study Design: single-centre, parallel-arms, PROBE (Prospective Randomized Open Blinded End-Point) trial.

The study will be submitted to the Ethical Committee of IRCCS NEUROMED and performed according to the Helsinki Declaration. All patients will sign an informed consent before inclusion into the study.

Inclusion criteria: patients with CLI (Rutherford classes 4, 5, 6), stenosis and/or complete occlusion of P3 popliteal artery segment, stenosis and/or complete occlusion of at least 1 leg vessel >40 mm in length, life-expectancy >12 months, possibility to perform angiogram at 12-months follow-up.

Exclusion criteria: life-expectancy <12 months, iodinated contrast media or paclitaxel allergy, impossibility to undergo dual antiplatelet therapy.

Randomization: Lesions will be randomly assigned to DEB PTA or standard PTA after successful passage of the guidewire. Randomization will be performed in blocks of 10 with the use of computer-generated random digits, and the assignments will be placed in sealed envelopes.

Intraoperative details:

PTA procedures are usually performed by an antegrade approach through a 5 Fr sheath, after systemic anticoagulation (Heparin Sodium 70 IU/kg). In patients randomised to DEB PTA, a predilatation with standard balloon is always performed. When more than 1 DEB is needed, a 5 mm overlapping zone between balloons is always considered. In all cases, regardless of type of balloon, inflation length is 3 minutes. At completion angiogram, in case of flow-limiting dissection or >30% residual stenosis, a further 3 minutes PTA is performed. Coronary stents are used as bailout.

Technical success is defined as the successful recanalization of target vessel with direct flow to the foot, with residual stenosis <30%. Inflow lesions of above-the-knee (ATK) segment are treated during the same session. Patients with bilateral lesions are treated in different procedures. After intervention, patients are usually treated with dual antiplatelet therapy (acetylsalicylic acid 100 mg/day and Clopidogrel 75 mg/day) for at least 4 weeks, followed by lifelong single antiplatelet therapy (acetylsalicylic acid 100 mg/day).

All DEB PTAs are performed by Ranger Balloon (Boston Scientific, Natick, MA, USA). This balloon is provided by Sterling platform associated with a loading tool aimed to protect the balloon surface during insertion inside the sheath, in order to avoid drug loss during intra-arterial navigation. Paclitaxel is coated to balloon surface by citrate ester in a peculiar form, allowing providing an optimal drug dose release at target vessel wall.

Follow-up: Duplex Ultrasound Scans (DUS) are scheduled at 1, 3 and 6 months from intervention. At 1 year follow-up, all patients undergo digital subtraction angiography (DSA). The latter DSA is compared with intraoperative diagnostic imaging using the same projections. Trophic lesions care is performed by weekly visits for the first 2 months, followed by bimonthly visits for the next 2 months. Visits are then scheduled monthly until ulcer healing. Planned minor amputations in non-infected patients are performed within 1 month from the index procedure.

Primary outcomes: 12-months binary restenosis rate, defined as lumen loss >50% at DSA.

Secondary outcomes: clinically driven target lesion revascularization (CD-TLR) rate, major amputations rate, wound healing rate, 12-months target vessel occlusion rate at DSA.

Acquired angiograms and DUS scans will be reviewed by 2 blinded investigators who will not actively participate in recruitment and will have no knowledge of randomization group.

Study power: Assuming a binary restenosis rate after conventional PTA of 75% and a reduction of at least 50% after DEB 4, a minimum of 41 lesions for group should be evaluated to have a statistical power of 90% and a significance level alpha=0.05 (two-sided).

Assuming a occlusion rate of target lesion after conventional PTA of 55% and a reduction of at least 60% after DEB 4, a minimum of 44 lesions for group should be evaluated to have a statistical power of 90% and a significance level alpha=0.05 (two-sided).

The number of lesions could be increased up to 50 for randomization group to maximise the power of the study.

Assuming a rate of eligible lesions per patient of 1.3, a minimum of 78 patients should be enrolled in the study.

Statistical analysis. Continuous variables will be expressed as means±standard deviation or medians with interquartile ranges and as percentage for categorical variables. Variables with positive skewness will be analysed after a logarithmic transformation.

To compare the characteristics of two randomization group, Student's t test will be used for continuous variables and X2 test for categorical variables (Exact Fisher's test will be used for cell with frequency <6).

Concordance data between ecodoppler and angiography will be tested by Bland-Altman method.

The "intention to treat" principle will be adopted for the analysis of the primary endpoints: the evaluation of efficacy takes into account the initial randomization independently from the compliance to the treatment of the subject.

The rate of primary outcomes between the two randomization group will be compared by Kaplan-Meier method, followed by long-rank test, e by multivariate logistic analysis, adjusted for possible confounding.

The data analysis will be generated using SAS/STAT software, Version 9.1.3 of the SAS System for Windows©2009. SAS Institute Inc. and SAS are registered trademarks of SAS Institute Inc., Cary, NC, USA.

Timeline:

Taking into account a recruitment capacity of our centre on 60 eligible patients per year, the recruitment phase will last 15 months for a total duration of the study of 36 months.

Month 0-3: protocol preparation, ethical committee approval, patient identification Month 4-19: enrolment of patients Month 12: ad interim analysis of results. Required because of the high rate of success of DEB reported by other studies.

Month 16-31: follow-up. Month 32-36: Data analysis and publication of results

ELIGIBILITY:
Inclusion Criteria:

* patients with CLI (Rutherford classes 4, 5, 6);
* stenosis and/or complete occlusion of P3 popliteal artery segment;
* stenosis and/or complete occlusion of at least 1 leg vessel >40 mm in length;
* life-expectancy >12 months;
* possibility to perform angiogram at 12-months follow-up.

Exclusion Criteria:

* life-expectancy <12 months;
* iodinated contrast media or paclitaxel allergy;
* impossibility to undergo dual antiplatelet therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
binary restenosis rate | 12-months
  binary restenosis rate has been defined as lumen loss >50% at DSA

SECONDARY OUTCOMES:
clinically driven target lesion revascularization (CD-TLR) rate | 12-months
major amputations rate | 12-months
wound healing rate | 12-months
target vessel occlusion rate | 12-months
  vessel occlusion rate at DSA

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Biello, MD, Principal Investigator — Neuromed IRCCS

REFERENCES:
- [Background] Forbes JF, Adam DJ, Bell J, Fowkes FG, Gillespie I, Raab GM, Ruckley CV, Bradbury AW; BASIL trial Participants. Bypass versus Angioplasty in Severe Ischaemia of the Leg (BASIL) trial: Health-related quality of life outcomes, resource utilization, and cost-effectiveness analysis. J Vasc Surg. 2010 May;51(5 Suppl):43S-51S. doi: 10.1016/j.jvs.2010.01.076. PMID 20435261
- [Background] Scheinert D, Duda S, Zeller T, Krankenberg H, Ricke J, Bosiers M, Tepe G, Naisbitt S, Rosenfield K. The LEVANT I (Lutonix paclitaxel-coated balloon for the prevention of femoropopliteal restenosis) trial for femoropopliteal revascularization: first-in-human randomized trial of low-dose drug-coated balloon versus uncoated balloon angioplasty. JACC Cardiovasc Interv. 2014 Jan;7(1):10-9. doi: 10.1016/j.jcin.2013.05.022. PMID 24456716
- [Background] Liistro F, Porto I, Angioli P, Grotti S, Ricci L, Ducci K, Falsini G, Ventoruzzo G, Turini F, Bellandi G, Bolognese L. Drug-eluting balloon in peripheral intervention for below the knee angioplasty evaluation (DEBATE-BTK): a randomized trial in diabetic patients with critical limb ischemia. Circulation. 2013 Aug 6;128(6):615-21. doi: 10.1161/CIRCULATIONAHA.113.001811. PMID 23797811
- [Background] Zeller T, Baumgartner I, Scheinert D, Brodmann M, Bosiers M, Micari A, Peeters P, Vermassen F, Landini M, Snead DB, Kent KC, Rocha-Singh KJ; IN.PACT DEEP Trial Investigators. Drug-eluting balloon versus standard balloon angioplasty for infrapopliteal arterial revascularization in critical limb ischemia: 12-month results from the IN.PACT DEEP randomized trial. J Am Coll Cardiol. 2014 Oct 14;64(15):1568-76. doi: 10.1016/j.jacc.2014.06.1198. PMID 25301459